CLINICAL TRIAL: NCT01469156
Title: Treatment of Polypoidal Choroidal Vasculopathy With High Dose Ranibizumab (Lucentis): A Phase I Safety Study.
Brief Title: Safety Study of 2.0mg Lucentis to Treat Polypoidal Choroidal Vasculopathy
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Southeast Retina Center, Georgia (Other)
Collaborators: Genentech, Inc. (Industry)
Responsible Party: Principal Investigator, Dennis M. Marcus, M.D., Dr. Dennis M. Marcus Principal Investigator, Southeast Retina Center, Georgia
Allocation: Randomized | Model: Single Group | Masking: Double | Purpose: Treatment
Other Study IDs: FVF4916s
Record Dates: First submitted 2011-11-03; First posted 2011-11-10 (Estimated); Results first posted 2022-12-12 (Actual); Last update posted 2022-12-12 (Actual); Status verified 2022-11

CONDITIONS: Polypoidal Choroidal Vasculopathy
Keywords: polypoidal choroidal vasculopathy; choroidal neovascularization; ranibizumab; Lucentis
MeSH Terms: conditions — Polypoidal Choroidal Vasculopathy; Choroidal Neovascularization | interventions — Ranibizumab

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- Ranibizumab 1.0 or 2.0 mg (HIGH DOSE) (Experimental): Intraocular injection of 1.0 or 2.0 mg/0.05 cc ranibizumab.
  Photodynamic therapy with visudyne or laser photocoagulation or intravitreal steroids may be considered as monotherapy or in combination with Ranibizumab at the investigator's discretion if rescue criteria are met
  Interventions: Drug: ranibizumab 0.5 or 2.0 mg/0.05 cc
- Ranibizumab 0.5 mg (Active Comparator): Intraocular injection of 0.5 mg/0.05 cc ranibizumab.
  Photodynamic therapy with visudyne or laser photocoagulation or intravitreal steroids may be considered as monotherapy or in combination with Ranibizumab at the investigator's discretion if rescue criteria are met
  Interventions: Drug: ranibizumab 0.5 or 2.0 mg/0.05 cc

INTERVENTIONS:
Drug: ranibizumab 0.5 or 2.0 mg/0.05 cc — ranibizumab (3:1 ratio of 2mg:0.5 mg ranibizumab) administered in three initial monthly doses followed by a 9 month period of criteria-based, as-needed retreatment and 12 month off drug safety follow up.
  Other Names: Lucentis

SUMMARY:
This Phase I/II study will investigate the safety and tolerability of intravitreally administered 0.5mg and 1.0 or 2.0mg Ranibizumab in three monthly doses followed by a 9 month period of criteria-based, as-needed retreatment and 12 month of drug safety follow up in subjects with exudative polypoidal choroidal vasculopathy (PCV) for a total of 24 months.

DETAILED DESCRIPTION:
Twenty eyes will be randomized will receive 3 consecutive monthly intravitreal 1.0 or 2.0 mg/0.5mg (3:1 ratio) Ranibizumab injection with the first injection occuring at Day 0 and second and third injection occuring at month 1 and month 2 respectively. Retreatment with intravitreal Ranibizumab or other therapies will be at the investigators discretion but guidelines for recommended retreatment.

ELIGIBILITY:
Inclusion Criteria:

* Males and Females >18 years of age. Females of child bearing potential will undergo urine pregnancy testing and be required to use appropriate methods of birth control.
* ICG and fluorescein angiographic characteristics consistent with active, leaking PCV with subfoveal lesions and/or subfoveal hemorrhage, lipid exudates, PED or fluid diagnosed within the past 6 months or diagnosed as newly active within the past 6 months. Subjects who completed the 24 month follow up in the original FVF3671s protocol may enter the study without necessarily demonstrating active exudative PCV at enrollment.
* Best-Corrected ETDRS Visual Acuity at 4 meters between 20/20 - 20/800.
* Lesion size - no limitations.
* Lesions Characteristics - leaking lesions consistent with PCV. No limitations on hemorrhage, fibrosis or atrophy.
* No therapy (includes non foveal laser, PDT, intravitreal steroids, TTT, radiotherapy, or anti-VEGF therapy) or intraocular surgery within the past 30 days for any condition.
* Clear ocular media to allow for photography/angiography.
* Ability to provide written informed consent and comply with study assessments for the full duration of the study.

Exclusion Criteria:

* Patients with features of age related macular degeneration such as abundant drusen and demographic features consistent with this diagnosis.
* Allergy to Fluorescein, ICG, Iodine, Shellfish.
* Pregnancy (positive pregnancy test)
* Any other condition that the investigator believes would pose a significant hazard to the subject if the investigational therapy were initiated.
* Participation in another simultaneous medical investigation or trial.
* Exclude other anti-VEGF agents as therapy options.
* History of previous subfoveal laser.
* Advanced glaucoma (IOP > 25 or cup/disc ration > 0.8)
* Any condition in the opinion of the investigator that would interfere with disease status/progression or jeopardize patients' participation in the study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2011-09; Primary Completion 2015-02 (Actual); Study Completion 2015-02 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Dennis M. Marcus, M.D., Principal Investigator — Southeast Retina Center
Locations (1):
- Southeast Retina Center, Augusta, Georgia, United States

RESULTS

PARTICIPANT FLOW:
Groups:
- Ranibizumab 1.0 or 2.0 mg (HIGH DOSE): Intraocular injection of 2.0 mg/0.05 cc ranibizumab or 1.0mg/0.05cc ranibizumab.
  Photodynamic therapy with visudyne or laser photocoagulation or intravitreal steroids may be considered as monotherapy or in combination with Ranibizumab at the investigator's discretion if rescue criteria are met
  ranibizumab 0.5 or 2.0 mg/0.05 cc: ranibizumab (3:1 ratio of 2mg:0.5 mg ranibizumab) administered in three initial monthly doses followed by a 9 month period of criteria-based, as-needed retreatment and 12 month off drug safety follow up.
- Ranibizumab 0.5 mg: Intraocular injection of 0.5 mg/0.05 cc ranibizumab.
  Photodynamic therapy with visudyne or laser photocoagulation or intravitreal steroids may be considered as monotherapy or in combination with Ranibizumab at the investigator's discretion if rescue criteria are met
  ranibizumab 0.5 or 2.0 mg/0.05 cc: ranibizumab (3:1 ratio of 2mg:0.5 mg ranibizumab) administered in three initial monthly doses followed by a 9 month period of criteria-based, as-needed retreatment and 12 month off drug safety follow up.
Period: Overall Study
Arm/Group | Ranibizumab 1.0 or 2.0 mg (HIGH DOSE) | Ranibizumab 0.5 mg
Started | 15 | 5
Completed | 15 | 5
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Ranibizumab 1.0 or 2.0 mg (HIGH DOSE): Intraocular injection of 2.0 mg/0.05 cc ranibizumab.
  Photodynamic therapy with visudyne or laser photocoagulation or intravitreal steroids may be considered as monotherapy or in combination with Ranibizumab at the investigator's discretion if rescue criteria are met
  ranibizumab 0.5 or 2.0 mg/0.05 cc: ranibizumab (3:1 ratio of 2mg:0.5 mg ranibizumab) administered in three initial monthly doses followed by a 9 month period of criteria-based, as-needed retreatment and 12 month off drug safety follow up.
- Total: Total of all reporting groups
Arm/Group | Ranibizumab 1.0 or 2.0 mg (HIGH DOSE) | Ranibizumab 0.5 mg | Total
Number analyzed (Participants) | 15 | 5 | 20
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 12 | 4 | 16
  >=65 years | 3 | 1 | 4
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 7 | 2 | 9
  Male | 8 | 3 | 11
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 0 | 0
  Not Hispanic or Latino | 15 | 5 | 20
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 1 | 0 | 1
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 7 | 1 | 8
  White | 7 | 4 | 11
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 15 | 5 | 20

OUTCOME MEASURES:

1. Primary Outcome: Incidence and Severity of Ocular and Systemic Adverse Events Will be Compared Between the 2.0mg or 1.0mg (HIGH DOSE) and 0.5 mg Groups.
Description: Examples include 30 letter loss, major subretinal hemorrhage, involving 75% or more clinical macula (arcade to arcade), disease related vitreous hemorrhage, injection-related endophthalmitis, retinal detachment, vitreous hemorrhage, study drug/procedure - related uveitis, incidence and severity of other adverse events, as identified by physical examination, subject reporting, and changes in vital signs.
Time Frame: 2 years
Measure: Number; unit: Adverse events
Groups:
- Control Group: Ranibizumab 0.5mg: standard-dose ranibizumab in 3 monthly loading doses, followed by 9 months of criteria-based, as-needed retreatment
- Ranibizumab 1.0mg or 2.0mg: high-dose ranibizumab in 3 monthly loading doses, followed by 9 months of criteria-based, as-needed retreatment
Arm/Group | Control Group: Ranibizumab 0.5mg | Ranibizumab 1.0mg or 2.0mg
Number analyzed (Participants) | 5 | 15
Adverse events
  Total Ocular and Notable Systemic AEs | 4 | 24
  Blurred or decreased vision | 0 | 6
  Floaters | 2 | 4
  Dark Spots | 0 | 3
  Injection site or ocular pain | 0 | 2
  Increased Cataracts | 0 | 2
  Subretinal hemorrhage | 0 | 1
  Superior hemorrhage | 0 | 1
  Increased Choroidal Neovascularization | 0 | 1
  Corneal abrasion | 0 | 1
  Trace epiretinal membrane | 0 | 1
  Flashes | 0 | 1
  Progression of edema | 0 | 1
  Light sensitivity | 1 | 0
  Elevated blood pressure | 1 | 0
Statistical Analysis 1: Comparison: Control Group: Ranibizumab 0.5mg vs Ranibizumab 1.0mg or 2.0mg; Purpose was to determine safety and efficacy of intravitreal high-dose ranibizumab in the treatment of active PCV; Test type: Other — Visually significant ocular or systemic AEs were predominantly mild or moderate. No significant safety signals were observed in either group.High- and standard-dose ranibizumab were generally well tolerated without evidence of ocular or systemic severe adverse events, including arterial thromboembolic events; p = 0.05, t-test, 2 sided — 28 ocular and non-ocular adverse events collected, in mild to moderate nature; data survey = 28, 95% CI 2-sided [0 to 28]; Visually significant ocular or systemic AEs that were either reported by subjects or identified by imaging and/or ocular exam

2. Secondary Outcome: Mean Best Corrected Visual Acuity Letter Change at 4 Meters Between Baseline and 12 Months
Time Frame: 12 months
Population: Randomized in a 3:1 ratio - number in participant flow is 20
Measure: Mean (Full Range); unit: letters
Groups:
- Ranibizumab 2.0 mg: Intraocular injection of 2.0 mg/0.05 cc ranibizumab.
  Photodynamic therapy with visudyne or laser photocoagulation or intravitreal steroids may be considered as monotherapy or in combination with Ranibizumab at the investigator's discretion if rescue criteria are met
  ranibizumab 0.5 or 2.0 mg/0.05 cc: ranibizumab (3:1 ratio of 2mg:0.5 mg ranibizumab) administered in three initial monthly doses followed by a 9 month period of criteria-based, as-needed retreatment and 12 month off drug safety follow up.
Arm/Group | Ranibizumab 2.0 mg | Ranibizumab 0.5 mg
Number analyzed (Participants) | 15 | 5
letters | 6.7 [-3 to 25] | -5 [-25 to 9]

3. Secondary Outcome: Change in Mean Central Foveal Thickness From Baseline
Time Frame: 12 Months
Population: Randomized in a 3:1 ratio
Measure: Mean (Standard Deviation); unit: um
Arm/Group | Ranibizumab 2.0 mg | Ranibizumab 0.5 mg
Number analyzed (Participants) | 15 | 5
um | -49.7 (100.71) | 94.4 (89.6)

4. Secondary Outcome: Mean Change From Baseline in Total Area of FA CNV Leakage Over 12 Months
Time Frame: 12 Months
Population: Randomized in a 3:1 ratio
Measure: Mean (Full Range); unit: mm^2
Arm/Group | Ranibizumab 2.0 mg | Ranibizumab 0.5 mg
Number analyzed (Participants) | 15 | 5
mm^2 | 2.38 [-1.12 to 8.71] | -0.38 [-1.12 to -0.02]

5. Secondary Outcome: Number of Participants at Month 3 With Best Corrected Visual Acuity Gain of 5, 10, and 15 or More Letters
Time Frame: 3 Months
Population: Randomized in a 3:1 ratio - number in participant flow is 20
Measure: Count of Participants; unit: Participants
Arm/Group | Ranibizumab 2.0 mg | Ranibizumab 0.5 mg
Number analyzed (Participants) | 15 | 5
Participants
  5-9 letters | 3 | 0
  10-14 letters | 2 | 0
  15 letters or more | 3 | 0
  Less than 5 letters | 6 | 0
  Unevaluable | 1 | 0

6. Secondary Outcome: Number of Participants at Month 6 With Best Corrected Visual Acuity Gain of 5, 10, and 15 or More Letters
Time Frame: 6 months
Population: Randomized in a 3:1 ratio - number in participant flow is 20
Measure: Count of Participants; unit: Participants
Arm/Group | Ranibizumab 2.0 mg | Ranibizumab 0.5 mg
Number analyzed (Participants) | 15 | 5
Participants
  5 letters | 3 | 1
  10 letters | 1 | 0
  15 or more letters | 4 | 0

7. Secondary Outcome: Number of Participants at Month 9 With Best Corrected Visual Acuity Gain of 5, 10, and 15 or More Letters
Time Frame: 9 Months
Population: Randomized in a 3:1 ratio - number in participant flow is 20
Measure: Count of Participants; unit: Participants
Arm/Group | Ranibizumab 2.0 mg | Ranibizumab 0.5 mg
Number analyzed (Participants) | 15 | 5
Participants
  5 letters | 3 | 0
  10 letters | 3 | 0
  15 letters | 2 | 0

8. Secondary Outcome: Number of Participants at Month 12 With Best Corrected Visual Acuity Gain of 5, 10, and 15 or More Letters
Time Frame: 12 Months
Population: Randomized in a 3:1 ratio - number in participant flow is 20
Measure: Count of Participants; unit: Participants
Arm/Group | Ranibizumab 2.0 mg | Ranibizumab 0.5 mg
Number analyzed (Participants) | 15 | 5
Participants
  5 letters | 4 | 1
  10 letters | 1 | 0
  15 letters | 3 | 0

9. Secondary Outcome: Mean Change Best Corrected Visual Acuity at 4 Meters at Baseline, Month 3, Month 6, Month 9, and Month 12
Time Frame: 12 months
Population: Randomized in a 3:1 ratio - number in participant flow is 20
Measure: Mean (Standard Deviation); unit: letters
Arm/Group | Ranibizumab 2.0 mg | Ranibizumab 0.5 mg
Number analyzed (Participants) | 15 | 5
letters
  Mean Change Baseline - M3 | 9.87 (15.27) | -2.8 (32.71)
  Mean Change Baseline - M6 | 10.23 (33.51) | -3.6 (2.35)
  Mean Change Baseline - M9 | 10.93 (43.81) | -6.8 (9.08)
  Mean Change Baseline - M12 | 6.37 (26.02) | -7.3 (20.11)

10. Secondary Outcome: Number of Participants at Month 3 With Best Corrected Visual Acuity Loss at 4 Meters of 5, 10 and 15 or More Letters
Time Frame: 3 months
Population: Randomized in a 3:1 ratio - number in participant flow is 20
Measure: Count of Participants; unit: Participants
Arm/Group | Ranibizumab 2.0 mg | Ranibizumab 0.5 mg
Number analyzed (Participants) | 15 | 5
Participants
  5 letters | 1 | 0
  10 letters | 0 | 0
  15 letters | 1 | 1

11. Secondary Outcome: Number of Participants at Month 6 With Best Corrected Visual Acuity Loss at 4 Meters of 5, 10 and 15 or More Letters
Time Frame: 6 months
Population: Randomized in a 3:1 ratio - number in participant flow is 20
Measure: Count of Participants; unit: Participants
Arm/Group | Ranibizumab 2.0 mg | Ranibizumab 0.5 mg
Number analyzed (Participants) | 15 | 5
Participants
  5 letters | 0 | 1
  10 letters | 0 | 1
  15 letters | 1 | 0

12. Secondary Outcome: Number of Participants at Month 9 With Best Corrected Visual Acuity Loss at 4 Meters of 5, 10 and 15 or More Letters
Time Frame: 9 months
Population: Randomized in a 3:1 ratio - number in participant flow is 20
Measure: Count of Participants; unit: Participants
Arm/Group | Ranibizumab 2.0 mg | Ranibizumab 0.5 mg
Number analyzed (Participants) | 15 | 5
Participants
  5 letters | 0 | 0
  10 letters | 0 | 0
  15 letters | 1 | 1

13. Secondary Outcome: Number of Participants at Month 12 With Best Corrected Visual Acuity Loss at 4 Meters of 5, 10 and 15 or More Letters
Time Frame: 12 months
Population: Randomized in a 3:1 ratio - number in participant flow is 20
Measure: Count of Participants; unit: Participants
Arm/Group | Ranibizumab 2.0 mg | Ranibizumab 0.5 mg
Number analyzed (Participants) | 15 | 5
Participants
  5 letters | 0 | 1
  10 letters | 0 | 0
  15 letters | 0 | 1

ADVERSE EVENTS:
Arm/Group | Control Group: Ranibizumab 0.5mg | Ranibizumab 1.0mg or 2.0mg
Serious Adverse Events (participants affected / at risk) | 0/5 | 0/15
Other Adverse Events (participants affected / at risk) | 2/5 | 9/15
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Control Group: Ranibizumab 0.5mg (N=5) | Ranibizumab 1.0mg or 2.0mg (N=15)
Affected vision (Eye disorders) | 1 (3) | 6 (14) — Blurred or decreased vision, floaters, dark spots, flashes, light sensitivity
Intravitreal injection side effects (Eye disorders) | 0 (0) | 2 (3) — Injection site or pain, subretinal hemorrhage
Increased cataract (Eye disorders) | 0 (0) | 2 (2) — Increased cataract from baseline measurement as determined during slit lamp ocular exam
Superior hemorrhage (Eye disorders) | 0 (0) | 1 (1) — Superior hemorrhage
Increased Choroidal neovascularization (Eye disorders) | 0 (0) | 1 (1) — As identified by FA
Corneal Abrasion (Eye disorders) | 0 (0) | 1 (1)
Trace epiretinal membrane (Eye disorders) | 0 (0) | 1 (1) — identified on clinical exam and OCT
Progression of edema (Cardiac disorders) | 0 (0) | 1 (1) — self reported by subject
Elevated Blood pressure (Cardiac disorders) | 1 (1) | 0 (0) — Self reported by subject

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2010-11-15): https://cdn.clinicaltrials.gov/large-docs/56/NCT01469156/Prot_SAP_000.pdf